CLINICAL TRIAL: NCT05432232
Title: The HistoSonics Investigational System for Treatment of Primary Solid Renal Tumors Using Histotripsy
Acronym: CAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HistoSonics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSP2276
Record Dates: First submitted 2022-06-17; First posted 2022-06-27 (Actual); Results first posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-10

CONDITIONS: Renal Cancer; Tumor, Solid; Kidney Cancer; Tumor; Tumor, Benign; Kidney Neoplasms
MeSH Terms: conditions — Kidney Neoplasms; Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a prospective, multi-center, single-arm, pilot trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- HistoSonics Investigational System (Experimental)
  Interventions: Device: HistoSonics Investigational System

INTERVENTIONS:
Device: HistoSonics Investigational System — The HistoSonics Investigational System is intended for the non-invasive destruction of kidney tissue using histotripsy, a non-thermal mechanical process of focused ultrasound.
  Other Names: Histotripsy

SUMMARY:
The purpose of this trial is to evaluate the technical success and safety profile of the HistoSonics Investigational System for the treatment of primary solid renal tumors.

DETAILED DESCRIPTION:
This trial is a prospective, multi-center, single-arm pilot trial designed to evaluate the effectiveness and safety profile of the HistoSonics Investigational System in treating primary solid renal tumors. Following histotripsy treatment of the solid renal tumor, subjects will undergo imaging ≤36 hours post-index procedure to determine technical success. Additionally, subjects will be followed 180 days (6 months) post-index procedure, with evaluations at the 14-day, 30-day, 90-day, and 180-day time points to establish the efficacy and safety profile of the HistoSonics Investigational System.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥18 years of age.
2. Subject has signed the Ethics Committee (EC) approved trial Informed Consent Form (ICF) prior to any trial related tests/procedures and is willing to comply with trial procedures and required follow-up assessments.
3. Subject is diagnosed with a non-metastatic solid renal mass ≤3cm confirmed via CT or MRI ≤ 30 days prior to the index procedure date.
4. Subject can tolerate general anesthesia.
5. Subject has an Eastern Cooperative Oncology Group Performance Status (ECOG PS) grade 0-2 at baseline screening.
6. Subject meets all the following functional criteria at ≤14 days prior to the planned index procedure date:

   * White Blood Cell (WBC) ≥3,000/mm3
   * Absolute Neutrophil Count (ANC) ≥1,200/mm3
   * Hemoglobin (Hgb) ≥9 g/dL
   * Platelet count ≥100,000/mm3 (≥100 10*9/L)
   * White Blood Cell (WBC) ≤40 cells/µL via urinalysis
   * Albumin ≤300,000 mg/L via urinalysis
7. Subject has an eGFR ≥45mL/min, ≤14 days prior to the planned index procedure date.
8. International Normalized Ratio (INR) score of <1.5:

   * If on anticoagulants, other than aspirin or non-steroidal anti-inflammatory drugs, assessment must be performed on the day of the procedure; OR
   * If only on aspirin or non-steroidal anti-inflammatory drugs, assessment must be performed ≤14 days prior to the planned index procedure date; OR
   * If not on anticoagulants, assessment must be performed ≤14 days prior to the planned index procedure date
9. Biopsy is required to determine the type of tumor and must be performed ≥14 days prior to the planned index procedure date.
10. The tumor selected for histotripsy treatment must be ≤3cm in longest diameter.
11. Subject has an adequate acoustic window to visualize targeted tumor using the HistoSonics Investigational System.
12. Subject will undergo histotripsy treatment of only one (1) tumor during the index procedure, regardless of how many tumors the subject has.

Exclusion Criteria:

1. Subject is pregnant or planning to become pregnant or nursing (lactating) during the trial period.
2. Subject is enrolled and being actively treated in another investigational pharmaceutical or device trial ≤30 days prior to planned index procedure date.
3. Subject is undergoing active chemotherapy for any cancer ≤14 days prior to planned index procedure date.
4. Subject is undergoing active immunotherapy ≤40 days prior to planned index procedure date.
5. In the Investigator's opinion, the subject has co-morbid disease(s) or condition(s) that would cause undue risk and preclude safe use of the HistoSonics Investigational System.
6. Subject is on dialysis or being considered for dialysis.
7. Subject has not recovered to Common Terminology Criteria for Adverse Events (CTCAE) grade 2 or better from any adverse effects (except alopecia and neuropathy) related to previous anti-cancer therapy.
8. Subject has an uncorrectable coagulopathy other than that induced by aspirin or non-steroidal anti-inflammatory drugs.
9. Subject has a planned cancer treatment (e.g., nephrectomy, chemotherapy, immunotherapy etc.) prior to completion of the 30-day follow-up visit.
10. Subject has had previous treatments with chemotherapy, radiotherapy, or both that have not been discontinued ≥14 days prior to the planned index procedure date and have not recovered (CTCAE grade 2 or better) from related toxicity (exclusive of alopecia and neuropathy).
11. Subject has previous treatment with immunotherapies that has not been discontinued ≥40-days prior to the planned index procedure date and has not recovered from related toxicity (CTCAE grade 2 or better).
12. Subject has a life expectancy less than one (< 1) year.
13. In the investigator's opinion, histotripsy is not a treatment option for the subject.
14. Subject has a concurrent condition that could jeopardize the safety of the subject or compliance with the protocol.
15. Subjects' targeted tumor has had prior locoregional therapy (e.g., ablation, embolization, radiation).
16. Subjects' tumor is not treatable by the HistoSonics Investigational System's working ranges (refer to User Guide).
17. In the physician's opinion, the anticipated risk of intervention outweighs the potential benefits of the intervention.
18. Subject has acute renal failure.
19. Subject has a genetic predisposition to kidney cancer such as:

    * Von Hippel Lindau (VHL)
    * Hereditary Papillary Renal Carcinoma (HPRC)
    * Birt-Hogg-Dubé Syndrome (BHD)
    * Tuberous Sclerosis Complex (TSC)
    * Hereditary Leiomyomata's Renal Cell Carcinoma (HLRCC)
    * Reed's Syndrome
    * Succinate Dehydrogenase B Deficiency (SDHB)
    * BRCA 1 associated protein -1 (BAP1) Renal Cell Carcinoma
    * MITF predisposed Renal Cell Carcinoma
20. Tumor is an angiomyolipoma.
21. Subject has a known sensitivity to contrast media and cannot be adequately pre-medicated.
22. The targeted tumor is not clearly visible with diagnostic ultrasound and either magnetic resonance imaging (MRI) or computerized tomography (CT).
23. Targeted tumor with adequate margin overlaps the renal pelvis, main renal vessel, ureter, or other vital structure.
24. Targeted tumor with adequate margin overlaps a non-targeted tumor visible via imaging.
25. The treatment of the tumor will not allow for an adequate margin as determined by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-03-23 (Actual); Primary Completion 2024-12-28 (Actual); Study Completion 2025-06-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds Teaching Hospitals NHS Trust, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wah TM, Abdel-Hadi O, Brandon J, Bhambra B, Glencross H, Occidental J, Stones JM, Vasudev N, Bhattarai S, Cartledge J. Early Clinical Histotripsy Treatment of Renal Cell Carcinoma. Cardiovasc Intervent Radiol. 2025 Jun;48(6):883-885. doi: 10.1007/s00270-025-04023-9. Epub 2025 Apr 28. No abstract available. PMID 40295402
- [Background] Wah TM, Amaral JF, Laeseke PF. Treatment of Primary Solid Renal Tumours Using Histotripsy: Study Protocol for the CAIN Feasibility Trial. Cardiovasc Intervent Radiol. 2025 Jun;48(6):857-865. doi: 10.1007/s00270-025-04035-5. Epub 2025 Apr 28. PMID 40295399

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial enrolled participants between March 2023 and November 2024 at one (1) UK site. All eligible subjects who provided informed consent were considered enrolled. Only subjects enrolled and treated with the HistoSonics Investigational System were assessed for the primary endpoints. Follow-up beyond 30 days was ongoing at the time of primary endpoint analysis.
Period: Participant Screening
Arm/Group | HistoSonics Investigational System
Started | 20
Screen Failures | 9
Completed | 11 (Eligibility criteria met and participant was eligible for treatment with histotripsy.)
Not Completed | 9
Period: Treatment to 30-Day Follow-up
Arm/Group | HistoSonics Investigational System
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Participants treated with histotripsy
Arm/Group | HistoSonics Investigational System
Number analyzed (Participants) | 11
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 71.0 [59.0 to 79.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 10
  Other | 1

OUTCOME MEASURES:

1. Primary Outcome: Primary Effectiveness: Technical Success
Description: Technical success, defined as complete coverage of the tumor as determined ≤36 hours post-index procedure by magnetic resonance imaging (MRI) or computerized tomography (CT). [Core Lab Adjudicated]
Time Frame: Up to 36 hours after the index procedure
Measure: Number (95% Confidence Interval); unit: percentage of tumors
Units Other Than Participants: tumors
Arm/Group | HistoSonics Investigational System
Number analyzed (Participants) | 11
Number analyzed (tumors) | 11
percentage of tumors | 100.0 [71.5 to 100.0]

2. Primary Outcome: Primary Safety: Freedom From Index Procedure Related Major Complications
Description: Freedom from index procedure related major complications, defined by Clavien-Dindo Classification Grade 3 or higher up to 30 days after the last histotripsy procedure. [Clinical Events Committee Adjudicated]
Time Frame: 30 days Post-Index Procedure
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HistoSonics Investigational System
Number analyzed (Participants) | 11
percentage of participants | 90.9 [58.7 to 99.8]

3. Secondary Outcome: Technique Efficacy (Primary)
Description: Percentage of targeted tumors successfully eradicated post-index procedure assessed via MRI or CT at 90-days post-index procedure without repeat Histotripsy [Core Lab Adjudicated]
Time Frame: 90 days Post-Index Procedure
Reporting Status: Not Posted, anticipated posting 2026-05

4. Secondary Outcome: Technique Efficacy (Secondary)
Description: Percentage of targeted tumors successfully eradicated post-index procedure assessed via MRI or CT at 90-days post-index procedure after repeat Histotripsy [Core Lab Adjudicated]
Time Frame: 90 days Post-Index Procedure
Reporting Status: Not Posted, anticipated posting 2026-05

ADVERSE EVENTS:
Time Frame: Histotripsy treatment through 30 days
Description: All adverse events reported starting at the time the participant was treated in the trial to the 30-day visit interval.
Arm/Group | HistoSonics Investigational System
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 3/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HistoSonics Investigational System (N=11)
Vomiting (Gastrointestinal disorders) | 1 (1)
Urinary retention postoperative (Injury, poisoning and procedural complications) | 1 (1)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HistoSonics Investigational System (N=11)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 3 (3)
Abdominal pain lower (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Intestinal dilatation (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Influenza like illness (General disorders) | 3 (3)
Pain (General disorders) | 2 (3)
Decreased appetite (General disorders) | 2 (2)
Pyrexia (General disorders) | 1 (1)
Upper aerodigestive tract infection (Infections and infestations) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1)
Procedural site reaction (Injury, poisoning and procedural complications) | 1 (1)
White blood cell count increased (Investigations) | 2 (2)
C-reactive protein increased (Investigations) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Headache (Nervous system disorders) | 2 (2)
Taste disorder (Nervous system disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 10 (10)
Flank pain (Renal and urinary disorders) | 2 (3)
Chromaturia (Renal and urinary disorders) | 1 (1)
Subcapsular renal haematoma (Renal and urinary disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoaesthesia (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-22): https://cdn.clinicaltrials.gov/large-docs/32/NCT05432232/Prot_SAP_000.pdf